CLINICAL TRIAL: NCT03415204
Title: Acupuncture for Post Operative Pain Following Total Knee or Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0104-17-ZIV
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2018-01

CONDITIONS: Arthroplasty Complications
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupuncture (Experimental)
  Interventions: Other: acupuncture
- no acupuncture (No Intervention)

INTERVENTIONS:
Other: acupuncture — acupuncture for post operative pain
  Arms: acupuncture

SUMMARY:
Post operative pain (POP) is a major obstacle on the road to healing, despite the increasing interest in postoperative pain management and development of pain control modalities (1). Postoperative pain is still insufficiently treated with more than 50% of patients suffering from moderate to severe pain early after surgery .Pain after orthopedic surgery is considered especially difficult to manage. Approximately half of total knee or hip arthroplasty patients present with extreme pain immediately after surgery. Total knee and hip arthroplasty often results not only in severe perioperative pain and debilitation, but chronic pain, joint stiffness, and functional disability many months or even years following the procedure. Various modalities of treating orthopedic POP exist, but the optimal management of postoperative pain remains controversial with no clear consensus of the best method.We suggest that acupuncture can be an effective treatment for post operative pain after total knee or hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent, above 18 years of age, about to undergo total knee or hip arthroplasty

Exclusion Criteria:

* Known mental disease, active cancer disease, coagulopathy, Hepatitis B,C.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
average post operative pain during time of hospitalization | average pain score during 5 days following operation
  post operative pain will measured twice daily - morning and afternoon during hospitalization time. patients will be asked to rate thier pain on a visual analog scale ranging from 0- no pain to 10 - severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel

REFERENCES:
- [Derived] Rubin L, Avraham Y, Sharabi-Nov A, Shebly T, Ben Natan M, Rothem DE. Acupuncture Effect on Analgesic Consumption and Cortisol Levels Following Total Knee Arthroplasty: A Randomized Controlled Trial. Med Acupunct. 2023 Oct 1;35(5):230-235. doi: 10.1089/acu.2023.0024. Epub 2023 Oct 17. PMID 37920858